CLINICAL TRIAL: NCT06628973
Title: Social Prescribing to Improve Adherence and Outcomes in Women With Heart Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Louise Pilote, Professor of Medicine, James McGill Chair, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-10346
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure; Cardiac Failure; Heart Decompensation; Congestive Heart Failure(CHF); Myocardial Failure
Keywords: Heart Failure; Social Determinants of Health; Adherence; Social Prescribing; Hospitalizations; Readmissions; Sex; Gender; Quality of Life; Congestive Heart Failure; Women
MeSH Terms: conditions — Heart Failure; Coitus

STUDY DESIGN:
Intervention Model Description: This study is an intention to treat, multicenter, open-labeled, randomized clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social prescription (Experimental): The intervention consists of SP, wherein patients identified as having significant SDOH-related vulnerabilities on the SPARK questionnaire or during an interview will have a consultation with a LW who will provide them with social prescriptions.
  Interventions: Behavioral: Social prescribing
- Control (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Social prescribing — The intervention consists of SP, wherein patients identified as having significant SDOH-related vulnerabilities on the SPARK questionnaire or during an interview will have a consultation with a LW who will provide them with social prescriptions. LWs are individuals who LINK individuals with social needs to existing community supports and services within the community
  Arms: Social prescription

SUMMARY:
Background: Heart Failure (HF) is the second most common cause of hospitalizations for women in North America. Non-adherence to guideline-directed medical therapy (GDMT) is associated with 50% of all treatment failures and high rates of hospitalizations and death. A recent Canadian study showed that adherence to three or more GDMT medications occurred in only 20% of Canadian HF patients. Despite clear guidelines on the pharmacologic management of HF and the introduction of new and effective drugs, adherence to GDMT in women with HF is low. Furthermore, the rates of hospitalizations have not improved in Canada over the last decade, and mortality in Canadian women with HF remains high. One explanation may be that social determinants of health (SDOH), which are known to be strong predictors of both adherence and adverse outcomes in HF, have not specifically been targeted to improve either adherence or outcomes in HF. Social prescribing (SP) is an innovative, non-medical intervention that aims to improve health by addressing SDOH. However, whether using SP to LINK clinical and social services for the benefit of socially vulnerable HF women can improve outcome is unknown. By targeting SDOH, which are strong predictors of adherence and outcomes in HF, and which have been shown to disproportionately disfavor women, SP has the potential to significantly improve medication adherence, quality of life and outcomes in women with HF.

Objectives: The overall aim of this study is to assess whether SP, through individualized, SDOH-targeted interventions, can improve adherence and quality of life in Canadian women with HF and at high risk for no adherence. Primary objective: To determine whether SP can improve adherence to GDMT. Secondary objective: To determine whether SP can improve quality of life.

Methods: This is an intention to treat, multicenter (five centers), and open-labeled, randomized clinical trial. Women with HF with two or more points on a weighted SDOH questionnaire (SPARK tool) will be randomly assigned to either SP or control group. Women in the SP group will meet with a link worker (LW) who will perform SP. SP will consist of personalized referrals to non-medical supports or services based on women's specific SDOH-related vulnerabilities and social needs. SP will address social needs such as issues with income, unemployment, transportation, mobility, dependents, housing, loneliness, mental health, health literacy, medication management and medical appointment schedules. Social prescriptions will be based on the interview conducted by the LW and will prioritize SDOH-related vulnerabilities identified on the SPARK questionnaire. Participants in the control group will receive standard care as is typically offered in the current specialized HF clinic in the participating centers. Controls will not meet with a LW, but, as usual, their physician or treating team may refer them to any specialists or services they deem necessary.

Outcome measures: The primary outcome will be adherence to GDMT measured with PDC obtained from provincial administrative databases and the secondary outcome will be quality of life measures including physical limitations, social limitations, as measured with the Kansas City Cardiomyopathy Questionnaire (KCCQ-12).

Sample size Calculations: The sample size was calculated using the primary outcome of adherence to GDMT measured with PDC as a continuous variable. In one observational study on adherence to HF medications which compared women and males adherence using PDCs, adherence in women was 63% with a SD of 23%. The impact of an absolute increase of 10% in PDC on clinical end points was considered significant. Using an alpha of 0.05 and a power of 0.80, a minimum of 166 participants would be needed to detect a statistically significant difference. Based on pilot data, the proportion of women followed in heart failure clinics is 28% and the proportion of eligible women (i.e. 1 point or more on the SPARK questionnaire) is about 30%. Considering a 30% refusal rate and a 5% dropout rate (intention to treat with registry based outcome), the five chosen centers should totalize 188 participants. The secondary outcome, the KCCQ, is a continuous variable for which a change of five points or more (5%) is considered clinically significant. Using an alpha of 0.05 and a power of 0.80, 126 patients would be required to detect such a difference.

Significance: SP holds immense potential for women with HF by addressing critical gaps in care. SP may help bridge the gap between healthcare providers and community resources, providing tailored support addressing SDOH that disproportionately affect women with HF. SP has the potential to significantly enhance adherence to GDMT, which has been shown to greatly, reduce hospitalizations and mortality in this vulnerable population.

DETAILED DESCRIPTION:
2. The Proposed Trial 2.1 Proposed Trial Design This study is an intention to treat, multicenter, open-labeled, randomized clinical trial. Patients will be matched within centers (i.e. compared to patients from the same center) to account for the different demographics of each center as well as regional and provincial particularities (see section 2.4). It will be conducted in five HF clinics, in five different Canadian hospitals from two provinces: Alberta and Quebec with whom collaborations have already been confirmed.

2.2 Trial Intervention The intervention has multiple phases: 1) preparation phase and LW selection, 2) LW training, 3) listing of community supports and services, 4) SP, 5) follow-up.

2.2.1 Preparation phase: The preparation phase of the trial will last six months and will, in part, be used to identify and train LW as well as to develop lists of available resources in the community for each center. Choosing appropriate LW will be an important part of the trial preparation. Link workers need to be highly motivated individuals who already have some knowledge of the communities served by the hospital. For instance, LW are often individuals who have already been working or volunteering in the community or the hospital. LW are typically not social workers since a LW should be "linking" and not doing social interventions per se.

2.2.2 LW training: The first goal of the training will be to teach LW how to assess and provide SP to vulnerable individuals. The training of LW will happen in three stages. The first step will be a series of online modules developed by the Alberta Healthy Aging group to train LW. The second will be a zoom-based bootcamp. We will leverage the expertise and resources of Dr. Alayne M. Adams, who serves as Co-Principal Investigator (Co-PI) and is an active member of the Canadian Social Prescribing Communities of Practice. Dr. Adams' extensive knowledge and access to numerous resources in the field of SP will be invaluable in structuring and organizing the boot camp. By tapping into Dr. Adams' expertise, we can ensure that the boot camp is well-designed and incorporates best practices in SP. This collaboration will enhance the effectiveness and impact of SP, ultimately benefiting the patients and communities involved. LWs will also be trained to find resources in communities they are not familiar with and to enter these resources in the project's databases. The third stage of the training will be longitudinal and consist of weekly virtual meetings between LW, PIs and the study coordinator. These meetings will provide continuous support for LW, updates and discussion about their patients. They will also be used to offer as needed training sessions based on needs that will arise. After the six months of preparation, these weekly meetings will continue throughout the intervention and data collection phases.

2.2.3 Listing of community supports and services: During the preparation phase, each LW will develop a unique list of community supports and services available in the areas they most serve. Resources identified will be indexed according to the population, needs and SDOH they are intended to address and entered into a database that will be regularly updated and accessible to the LW to search as needed.

As the participating hospitals will be referral centers, patients will come from communities often far from the hospital and, therefore, resources will be numerous and spread out. Part of the training for LWs will be to teach them to use existing databases and individuals in the community who can help identify resources not already indexed on the web platform. Each new resource identified will then be indexed so that a more comprehensive database is built over time and available afterward. Resources commonly available in the community are patient support groups, subsidized or volunteer transportation services, food banks, housing support, employment support, physical activity groups, social work in the community and associations to support immigrants and allophones.

2.2.4 SP: The intervention consists of SP, wherein patients identified as having significant SDOH-related vulnerabilities on the SPARK questionnaire or during an interview will have a consultation with a LW who will provide them with social prescriptions. LWs are individuals who LINK individuals with social needs to existing community supports and services within the community (Appendix 6). During these consultations, the LW will engage with patients to understand their individual needs using a structured interview which includes the SPARK questionnaire. Based on this assessment, the LW will then perform SP consisting of written, individualized social prescriptions (i.e. referrals to existing community supports and service) to address their SDOH-related vulnerabilities and social needs. SP can help address needs such as low income, unemployment, transportation, mobility, dependents, housing, loneliness, mental health, health literacy, medication management and medical appointments schedule. Consultations will take place in specialized HF clinic.

At the time of the prescribing, many resources available in the community will have already been indexed by keywords on a database during the first phase of the trial (see above) and available to the LW to search. SDOH from the SPARK questionnaire will be part of the keywords used for the indexation and will be directly searchable on the platform (described in 2.2.3).

2.2.5 Follow-up: Structured follow-up calls will be made at seven and fourteen days after the initial prescription and then, monthly, or as needed based on social needs thereafter. Follow-up calls will serve two purposes. First, they will be used to assess if the patient has engaged in the activities prescribed and whether the activities fulfill their intended purpose. Second, they will assess whether patients' needs have changed since previous contact. When indicated, new social prescriptions will be provided.

Participants in the control group will receive standard of care as is typically offered in the current specialized HF clinic in participating centers. Controls will meet, as usual, with their physician or treating team who may refer them to any specialists or services they deem necessary. Follow-up time and measurements are the same in both the intervention and control arm.

2.3 Proposed practical arrangements for allocating participants to trial arms Participants will be first assessed using the SPARK questionnaire. Participants with a score of two or more points will then be randomly allocated in a 1:1 ratio to either SP or control arm.

2.4 Methods for Protecting Against Risk of Bias At the analysis stage, patient will be matched within centers (i.e. only compared to patients from the same center) to account for the different demographics of each center as well as regional and provincial particularities treating different types of populations. To limit the effect of survivorship bias on the secondary PROs measured with the KCCQ, they will be measured at six months and one year. Blinding for physicians in this study is not possible given the intervention will occur in the clinic, where it is likely to be noticed. Similarly, we cannot ask participants to hide the intervention from their treating team. Furthermore, our secondary outcome, the KCCQ, will be administered by LW who cannot be blinded to the intervention.

2.5 Inclusion and Exclusion Criteria Participants will be included in the study if they are (1) women, (2) 18 years of age or older, (3) have documented HF of any etiology, (4) have valid personal health identifier, (5) have two or more points on the weighted SPARK questionnaire. Patients not meeting inclusion criteria, who do not take HF medications, who are not residents of the province where they are being followed or who have opted out from their provincial health registry will be excluded. Patients with severe cognitive impairment or other conditions that significantly impact the ability to participate in SP will also be excluded.

2.6 Proposed Duration of Intervention Period (1 year) The recruitment and intervention period will last 1 year and the duration of the intervention by the LW will span 1 year (see Gantt chart in Appendix 4).

2.7 Proposed Duration of Follow-Up (1 year) For both primary and secondary outcomes, the proposed duration of follow-up after initial intervention is 1 year.

2.8 Proposed Primary and Secondary Outcomes The primary outcome will be the adherence to GDMT measured with the proportion of days covered (PDC). PDC(59), calculated as the sum of the number of unique days during which the patient had medication available, divided by a fixed time interval of 6-, or 12-months as applicable. The resulting ratio provides an estimate of the proportion of time the patient had access to their medication.

The secondary outcome will be the KCCQ overall score. The KCCQ encompasses the following relevant PROs: physical limitations, social limitations, symptoms and QoL. It will be administered three times, at baseline, six months and one year after the initial intervention. The validity of the KCCQ has been tested in diverse clinical settings and etiologies of HF(30, 60, 61). The KCCQ score ranges from 0 to 100 and is often divided into quartiles with 0 to 25 being very poor to poor, 26 to 49 being poor to fair, 50 to 74 being fair to good, and 75 to 100 being good to excellent(62). For this project we will be using the short form of the KCCQ which is simple and more convenient and has shown excellent correlation with the original questionnaire(63).

2.9 Outcome Measures PDC will be obtained by accessing provincial administrative health records. We will be using PDC as a continuous variable, and a significant change in adherence will be defined as a 10% difference based on findings from previous studies(64). GDMT medications include beta-blockers, angiotensin-converting enzyme inhibitors, angiotensin receptor blockers, angiotensin receptor, neprilysin inhibitors, sodium-glucose transport protein 2 (SGLT2) inhibitors and mineralocorticoid receptor antagonists(65). GDMT medications evaluated for adherence will be the ones prescribed at baseline or at any time during the follow-up period of 1 year. We will also obtain historical PDC data to adjust for PDC rates at baseline in the two groups. The KCCQ will be filled by LW for patients randomized to the SP and controls as well.

2.10 Sample Size Calculations The sample size was calculated based on the primary outcome of adherence to GDMT using PDC, a continuous variable. In one observational study on adherence to HF medications which compared women and males adherence using PDC, adherence in women was 63% with a SD of 23%(64). Increase of 10% increase in PDC on clinical end points was considered significant(64). Therefore, using an alpha of 0.05 and a power of 0.80, a minimum of 166 participants would be needed to detect such a difference.

Based on pilot data (Appendix 5), the proportion of women followed in heart failure clinics is about 28% and the proportion of eligible women (i.e. two or more points on the SPARK questionnaire) is about 30%. Considering a 30% refusal rate and a 5% dropout rate (intention to treat with registry based outcome), the five chosen centers should totalize 188 participants.

The secondary outcome, the KCCQ, is also a continuous variable for which a change of five points or more (5%) is considered clinically significant(66-68). Using an alpha of 0.05 and a power of 0.80, a total of 126 patients would be required to detect such a difference which is within the above sample size.

2.11 Health Economics and QoL measures Health economics will not be addressed in this project. QoL measures will be measured with the KCCQ and are the secondary outcome of this project, as detailed above.

2.12 Recruitment To better identify women patients with HF vulnerable to nonadherence, we will utilize the SPARK questionnaire that will be administered during patient visits to the clinic. This evidence-based instrument is aimed at integrating social determinants data with clinical data. The SPARK tool will be implemented in our clinics, and we will construct an intuitive database platform tailored for SDOH data collection. Tools will be implemented via paper or electronic form. Instruction will be included, and it will be user-friendly without the need for external assistance. Participants from centers randomized to the intervention, with two points or more on the SPARK questionnaire, meaning at least a moderate (two points) increase in the risk of non-adherence and adverse outcomes, will be referred to the LW for SP.

The SPARK questionnaire has not previously been used to identify patients at higher risk of nonadherence. Each element of the SPARK questionnaire will be weighted using a point system: one point for elements associated with a small increase in the risk of non-adherence, two points for elements associated with a moderate risk increase and three points for elements associated with a high-risk increase.

Rate of enrollment: Based on preliminary data from McGill University Health Center (MUHC) HF clinic, it is assumed that each centre will be able to contribute an average of 50 women participants for a total of 250 patients during the one year.

2.13 Compliance Adherence to HF medications is our primary outcome and will be measured using PDC detailed above. Adherence to the initial SP, i.e. the first interview with the LW, is expected to be very high as participants will have consented to meet the LW only a few minutes before the interview. Adherence to social prescriptions is expected to be lower and will be measured during the structured follow-up calls made by LW and will constitute an important result of this project. Very limited quantitative data exists with regards to adherence to social prescriptions. In one study, adherence to social services was increased by 15% in the SP group when compared to a self-referred group (48% vs 33%, p<0.01). In qualitative studies, the relationship and trust with the LW has been repeatedly identified as a strong driver of adherence to SP.

2.14 Loss to Follow-Up Follow-up assessments will occur in person between participants and LW during in-person clinical appointments or more often virtually, via email or telephone, based on the participant's preference in both groups. Reasons for non-participation and dropout will be tracked.

2.15 Number of Centres Involved We have confirmed collaboration with our five participating centers. In the province of Quebec. We have three centers in the Montreal area: 1) McGill University Health Center Hospitals - Royal Victoria Hospital (Abinav Sharma) and 2) Montreal General Hospital (Thao Huynh); 3) Montreal Heart Institute (Anique Ducharme). In the province of Alberta, we have two hospitals in Edmonton: 1) Heart Function Clinic (Gavin Y. Oudit) and 2) CKHUi heart centre (Marc Benoit).

2.16 Analyses Descriptive Analyses: A CONSORT flow chart will be created to outline patients' enrolment. The clinical and demographic characteristics of the study participants, including age, comorbidities, SDOH and social vulnerability levels based on the SPARK questionnaire will be collected. Social prescriptions will also be described.

Main Analyses: Both primary outcome and secondary outcomes will be compared between the SP and control arms using multivariate linear regression models adjusted for relevant clinical variables and SDOH. Participants will be matched within centers (i.e. compared to participants from the same center only) to account for centers following different types of patients.

Secondary Outcomes: The secondary outcome will be the KCCQ scores. Scores will be compared between SP and control arms using multivariate linear regression models adjusted for relevant clinical variables and SDOH.

2.17 Frequency of Analyses Analyses will be only performed once, at the end of follow-up at 1 year after the last patient has been enrolled.

2.18 Subgroup Analyses The different components of the SPARK questionnaire will allow for numerous subgroup analyses. Notably, we will look at different races, income tertials and education. From patient's file we will also be able to look specifically at patients with diseases associated with worse SDOH such as diabetes and chronic kidney disease. We also plan to look secondary outcomes such as hospitalizations and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18 years of age or older
* Documented HF of any etiology
* Valid personal health identifier
* Two or more points on the weighted SPARK questionnaire

Exclusion Criteria:

* Patients not meeting inclusion criteria
* Do not take HF medications
* Not residents of the province where they are being followed or who have opted out from their provincial health registry
* Patients with severe cognitive impairment or other conditions that significantly impact the ability to participate in SP will also be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of days | 6- 12 months
  The primary outcome will be the adherence to GDMT measured with the proportion of days covered (PDC). PDC(59), calculated as the sum of the number of unique days during which the patient had medication available, divided by a fixed time interval of 6-, or 12-months as applicable. The resulting ratio provides an estimate of the proportion of time the patient had access to their medication

SECONDARY OUTCOMES:
KCCQ overall score | 12 months
  The KCCQ encompasses the following relevant PROs: physical limitations, social limitations, symptoms and QoL. It will be administered three times, at baseline, six months and one year after the initial intervention. The validity of the KCCQ has been tested in diverse clinical settings and etiologies of HF. The KCCQ score ranges from 0 to 100 and is often divided into quartiles with 0 to 25 being very poor to poor, 26 to 49 being poor to fair, 50 to 74 being fair to good, and 75 to 100 being good to excellent. For this project we will be using the short form of the KCCQ which is simple and more convenient and has shown excellent correlation with the original questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of the McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
For ethical reasons we cannot share participants personal information